CLINICAL TRIAL: NCT06367868
Title: Evaluation of the Effect of Cerebrospinal Fluid Drainage on Optic Nerve Sheath Diameter in Patients Installed External Ventricular Drainage Catheter Due to Intracranial Pathology in the Intensive Care Unit
Brief Title: Optic Nerve Sheath Diameter: A Non-Invasive Indicator of Intracranial Pressure in the Intensive Care Unit Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gülşah ORAK, Medical Doctor-Anesthesiology and Reanimation, Istanbul University - Cerrahpasa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: E-83045809-604.01.02-179951
Record Dates: First submitted 2024-04-05; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: ICP (Intracranial Pressure) Increase; Optic Nerve Sheath Diameter; Intracranial Hypertension
Keywords: ONSD; ultrasonography; noninvasive; increased intracranial pressure
MeSH Terms: conditions — Intracranial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Before Drainage (Experimental): Optic nerve sheath diameter and intracranial pressure will be measured before CSF drainage
  Interventions: Procedure: After 5 ml CSF Drainage

INTERVENTIONS:
Procedure: After 5 ml CSF Drainage — Optic Nerve Sheath Diameter and Intracranial Pressure measurements will be after 5 ml CSF drainage

SUMMARY:
Determination of high intracranial pressure (ICP) is necessary for the treatment of patients with raised ICP to improve long-term neurological outcomes. Ultrasonographic optic nerve sheath diameter (ONSD) measurement is a noninvasive, easily performed and cost effective technique for detecting high ICP.

DETAILED DESCRIPTION:
ICP measurements via ventricular catheters provide CSF drainage and ICP reduction. The normal ICP value is less than 15 mmHg in adults. In the literature the correlation of ONSD and invasive ICP measurements were determined. The aim of study is to evaluate the correlation of ONSD and direct ICP measurements and to determine cut off ONSD value to detect ICP ≥15 mmHg.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 aged patients
* With an external ventricular drainage catheter due to intracranial pathology

Exclusion Criteria:

* Under the age of 18
* Orbital tumors
* Graves' disease
* Exophthalmos
* Sarcoidosis
* Optic neuropathy
* Meningitis
* Ocular trauma
* Lung diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Intracranial Pressure-1 (ICP-1) | baseline time
  Measurement of intracranial pressure before cerebrospinal fluid (CSF) drainage
Optic Nerve Sheath Diameter-1 (ONSD-1) | baseline time
  Measurement of optic nerve sheath diameter before cerebrospinal fluid drainage

SECONDARY OUTCOMES:
Intracranial Pressure-2 (ICP-2) | 2 minutes after CSF drainage
  Measurement of intracranial pressure 2 minutes after cerebrospinal fluid (CSF) drainage
Optic Nerve Sheath Diameter-2 (ONSD-2) | 2 minutes after CSF drainage
  Measurement of optic nerve sheath diameter 2 minutes after cerebrospinal fluid drainage

CONTACTS AND LOCATIONS:
Overall Officials: GULSAH ORAK, Study Director — Istanbul University - Cerrahpasa; OZLEM KORKMAZ DİLMEN, Study Chair — Istanbul University - Cerrahpasa; EREN FATMA AKCİL, Study Chair — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Fatıh, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Robba C, Santori G, Czosnyka M, Corradi F, Bragazzi N, Padayachy L, Taccone FS, Citerio G. Optic nerve sheath diameter measured sonographically as non-invasive estimator of intracranial pressure: a systematic review and meta-analysis. Intensive Care Med. 2018 Aug;44(8):1284-1294. doi: 10.1007/s00134-018-5305-7. Epub 2018 Jul 17. PMID 30019201
- [Background] Muller SJ, Henkes E, Gounis MJ, Felber S, Ganslandt O, Henkes H. Non-Invasive Intracranial Pressure Monitoring. J Clin Med. 2023 Mar 13;12(6):2209. doi: 10.3390/jcm12062209. PMID 36983213
- [Background] Sharawat IK, Kasinathan A, Bansal A, Sahu JK, Sodhi KS, Dogra MR, Sankhyan N. Evaluation of Optic Nerve Sheath Diameter and Transcranial Doppler As Noninvasive Tools to Detect Raised Intracranial Pressure in Children. Pediatr Crit Care Med. 2020 Nov;21(11):959-965. doi: 10.1097/PCC.0000000000002523. PMID 32852360
- [Background] Kimberly HH, Shah S, Marill K, Noble V. Correlation of optic nerve sheath diameter with direct measurement of intracranial pressure. Acad Emerg Med. 2008 Feb;15(2):201-4. doi: 10.1111/j.1553-2712.2007.00031.x. PMID 18275454